CLINICAL TRIAL: NCT05531734
Title: MONITORING OF ATTENTION ACCORDING TO FATIGUE IN THE HEALTHY SUBJECT
Acronym: MOTIVATES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP220576; 2022-A01959-34 (Other: IDRCB)
Record Dates: First submitted 2022-06-14; First posted 2022-09-08 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: FATIGUE; Sleep Deprivation
Keywords: Measurement tool; EEG data; sleep deprivation; attention; electroencephalogram
MeSH Terms: conditions — Fatigue; Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- volunteers (Experimental): Health volunteers
  Interventions: Device: NaoX Intra-Auricular Device (IAD) monitoring EEG data; Behavioral: Simple psychometric tests

INTERVENTIONS:
Device: NaoX Intra-Auricular Device (IAD) monitoring EEG data — Intrauaricular measurement tool developed by NaoX Technology to retrieve EEG type data.
Behavioral: Simple psychometric tests — Associated with simple and self-managed psychometric tests.

SUMMARY:
To develop an easy-to-use measurement tool for monitoring fatigue and alertness, particularly in sleep-deprived subjects.

DETAILED DESCRIPTION:
Objective and primary endpoint:

Demonstrate that the NaoX measurement tool detects sleep deprivation in medical residents performing medical shifts.

The primary endpoint is the detection of a significant decrease in Coefficient Alpha Attenuation (CAA) between the pre- and post-sleep deprivation measurements.

The data analysis will be blinded to the measurement.

Secondary endpoints and objectives :

Demonstrate a link between the Alpha Attenuation Coefficient (AAC) measured by the NaoX measurement tool and the vigilance tests.

Endpoint: significant increase in PVT (Psychomotor Vigilance Task) time associated with a significant decrease in Alpha Attenuation Coefficient (AAC).

Demonstrate a link between the Alpha Attenuation Coefficient (AAC) measured by the NaoX measurement tool and the state of fatigue experienced.

Endpoint: significant increase in Karolinska Sleepiness Scale (KSS) score associated with a significant decrease in Alpha Attenuation Coefficient (AAC).

Experimental scheme:

3 cycles of 2 recordings with the NaoX measurement tool associated with a self-questionnaire and vigilance tests (approximately 30 minutes per recording), carried out before and after a night shift by a medical resident.

Population targeted:

Medical residents performing night shifts of at least 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers.
* Male, female.
* Medical residents.
* Aged between 24 and 34 years.
* Doing emergency, intensive care or "inside" shifts.
* Working in a health institution.
* No history of epilepsy.
* No background treatment that could have an impact on the EEG (electroencephalogram) data (type: benzodiazepines, anti-epileptics).
* No significant change in background treatment during the study, if any.
* Affiliation to the social security system.
* Informed volunteer who has signed a consent form.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
EEG data collected by head phone like EEG electrodes developed by NaoX Technologies | through study completion, an average of 12 hours
  Demonstrate that the NaoX head phone like EEG electrodes detects sleep deprivation in medical residents performing medical shifts.
  The primary endpoint is the detection of a significant decrease in Coefficient Alpha Attenuation (CAA) between the pre- and post-sleep deprivation measurements.
  The data analysis will be blinded to the measurement.

SECONDARY OUTCOMES:
Demonstrate a link between the Alpha Attenuation Coefficient (AAC) measured by NaoX head phone like EEG electrodes and the vigilance tests | through study completion, an average of 12 hours
  Endpoint: significant increase in PVT (Psychomotor Vigilance Task) time associated with a significant decrease in Alpha Attenuation Coefficient (AAC).
Demonstrate a link between the Alpha Attenuation Coefficient (AAC) measured by the NaoX head phone like EEG electrodes tool and the state of fatigue experienced | through study completion, an average of 12 hours
  Endpoint: significant increase in Karolinska Sleepiness Scale (KSS) score associated with a significant decrease in Alpha Attenuation Coefficient (AAC).

CONTACTS AND LOCATIONS:
Overall Officials: Jean BERGOUNIOUX, MD, PhD, Principal Investigator — Pediatric Intensive Care Unit, Raymond Poincaré Hospital, APHP
Locations (1):
- Pediatric Intensive Care Unit, Raymond Poincaré Hospital, APHP, Garches, France

IPD SHARING:
Plan to Share IPD: No